CLINICAL TRIAL: NCT06111274
Title: A Multicenter, Open-Label Phase II Study To Evaluate The Efficacy And Safety Of ABSK021 In Combination With Chemotherapy With Or Without Toripalimab In Patients With Advanced Pancreatic Cancer
Brief Title: A Phase 2 Study of ABSK021 in Patients With Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK021-202
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABSK021 with chemotherapy (Experimental): There are 2 cohorts in both part A and Part B. In cohort 1, the participant will receive the treatment of ABSK021 in combination with chemotherapy (the Gemcitabine and nab-Pacilitaxel) , 3 weeks as one cycle, about 8 cycles in total.
  Interventions: Drug: Pimicotinib (ABSK021)
- ABSK021 in combination with chemotherapy plus the Toripalimab (Experimental): There are 2 cohorts in both part A and Part B. In cohort 2, the participant will receive the treatment of ABSK021 in combination with chemotherapy (the Gemcitabine and nab-Pacilitaxel), with Toripalimab, 3 weeks as one cycle, about 8 cycles in total.
  Interventions: Drug: Pimicotinib (ABSK021)

INTERVENTIONS:
Drug: Pimicotinib (ABSK021) — The ABSK021 will be taken orally, once daily; The Gemcitabine and nab-Pacilitaxel will be administrated with intravenous infusion on day 1 and 8 of each cycle; The Toripalimab will be administrated with intravenous infusion on day 1 of each cycle.
  Other Names: Gemcitabine; nab-Pacilitaxel; Toripalimab

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of Pimicotinib (ABSK021) in combination with chemotherapy with or without Toripalimab in patients with advanced pancreatic cancer. The main questions it aims to answer are:

* Whether the Pimicotinib (ABSK021) in combination with chemotherapy with or without Toripalimab is safe in patients with advanced pancreatic cancer.
* Whether the Pimicotinib (ABSK021) in combination with chemotherapy with or without Toripalimab is effective in patients with advanced pancreatic cancer.

Participants will be asked to complete the study procedures:

* Receive the administration of Pimicotinib (ABSK021) in combination with chemotherapy with or without Toripalimab about 24 weeks in study Part A or Part B.
* Receive the administration of Pimicotinib(ABSK021) about 24 weeks in study part 2.
* Complete the study procedures specified in the protocol, which is guided by researchers.

DETAILED DESCRIPTION:
This is a phase II, open-label study to evaluate safety, tolerability, pharmacokinetics (PK), and clinical benefit of Pimicotinib (ABSK021) in combination with chemotherapy with or without Toripalimab in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-75 years old. The subjects must have informed consent to the study, and signed the written informed consent voluntarily.
* Diagnosis as non resectable local advanced or metastatic pancreatic cancer by histology or cytology.
* Measurable disease as defined by RECIST 1.1.
* Without systemic treatment for pancreatic cancer.
* ECOG physical strength score 0-2
* Estimated survival time >=3 months.
* The adequate bone marrow fuction and coagulation function

Exclusion Criteria:

* Known allergy or hypersensitivity to any components of the investigational drug product.
* Previous treatment with highly selective inhibitors targeting Colony Stimulating Factor 1 (CSF-1)/Colony Stimulating Factor 1 Receptor (CSF-1R).
* With Breast Cancer Gene 1/2 (BRCA1/2) gene mutation.
* With a history of other malignancies within 5 years.
* During the trial, other chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy (except for local symptomatic radiotherapy) or traditional Chinese medicine must be used for anti-tumor treatment.
* With conditions that significantly affected the absorption of oral drug.
* Surgical treatment is required within 4 weeks before the first administration, or unhealed, infected, or dehiscence of previous surgical wounds.
* During the 2 weeks prior to the first administration of this study, the patient was receiving chronic systemic steroid treatment or any other form of immunosuppressive treatment.
* Concomitant use of strong inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4) within 14 days prior to randomization.
* Previous peripheral neuropathy > grade 1 (Common Terminology Criteria for Adverse Events, version 5.0).
* Diagnosed with immune deficiency or interstitial lung disease.
* The patients were vaccinated within 4 weeks before the first treatment.
* Participated in any drug clinical trial within 4 weeks before the first treatment.
* Active central nervous system (CNS) metastases.
* Impaired cardiac function or clinically significant cardiac disease.
* Known active liver or biliary disease, or other diseases that may lead to abnormal liver function test results during the study.
* Known active infections from certain viruses, bacteria or parasites.
* Patients with refractory/uncontrolled ascites or pleural effusion.
* Pregnant or lactating women.
* Any other clinically significant comorbidities, which in the judgment of the Investigator, should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Safety Event Occurance | From the day signed informed consent form to day 90 after the end of cycle 8 (each cycle is 21 days)
  The Number of Participants With Adverse Event (AE), a Serious Adverse Event (SAE) and Dose Limiting Toxicities (DLT) Event.
Objective Response Rate (ORR) | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  The Percentage of Participants with confirmed Complete Response and Partial Response, in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)

SECONDARY OUTCOMES:
Duration of Response | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  Duration of response (DOR) is defined as the time from the date of the first documentation of confirmed response (Complete Response or Partial Response) to the first objective documentation of progressive disease (PD) per RECIST v1.1 per Investigator assessment, or to death due to any cause in the absence of documented PD.
Progression Free Survival | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  Progression-free survival (PFS) was defined as as the time from the first dose to the first objectively documented disease progression per RECIST v1.1 per Investigator assessment, or death due to any cause in the absence of documented progressive disease (PD). PFS was analyzed using Kaplan-Meier methods.
Overall Survival | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  Overall survival (OS) was defined as the time from first dose of study drug to death due to any cause. OS was calculated using the Kaplan-Meier method.
The exposure of ABSK021 | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  The Area Under the Concentration Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) Normalized by Dose.
The Maximum Concentration of ABSK021 | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  Maximum Observed Concentration (Cmax)
The Minimum Concentration of ABSK021 | From the cycle 1 day 1 to the end of cycle 8 (each cycle is 21 days)
  Minimum Observed Concentration (Cmin)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Shanghai East Hospital Tongji University, Shanghai
  - Union Hospital Tongji Medical College Huazhong University of science and technolog, Wuhan

IPD SHARING:
Plan to Share IPD: No